CLINICAL TRIAL: NCT06859879
Title: A Combined Supplementation of Rosemary and Daylily for Enhancing Sleep Quality in Middle-Aged Adults
Acronym: RESTORE-ENG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Principal Investigator, Sergej Ostojic, Professor, University of Novi Sad, Faculty of Sport and Physical Education
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 51-02-18
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Sleep
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental 1: Low-dose (Experimental): One capsule of active Rosemary and Daylily extract and one placebo capsule
  Interventions: Dietary Supplement: Dietary Supplement: low-dose Rosemary and Daylily extract
- Experimental 2: Medium-dose (Experimental): Two capsules of active Rosemary and Daylily extract
  Interventions: Dietary Supplement: Dietary Supplement: medium-dose Rosemary and Daylily extract
- Experimental 3: Control (Placebo Comparator): Two capsules of placebo
  Interventions: Dietary Supplement: Dietary Supplement: control

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: low-dose Rosemary and Daylily extract — Supplement containing Rosemary and Daylily extract
  Arms: Experimental 1: Low-dose
Dietary Supplement: Dietary Supplement: medium-dose Rosemary and Daylily extract — Supplement containing Rosemary and Daylily extract
  Arms: Experimental 2: Medium-dose
Dietary Supplement: Dietary Supplement: control — Supplement containing placebo
  Arms: Experimental 3: Control

SUMMARY:
This study aims to investigate the impact of supplementation with two different doses of Rosemary and Daylily herbal extract on various health outcomes in middle-aged adults. Over an eight-week period, the trial will assess improvements in sleep quality, circadian rhythms, energy metabolism, and relevant biochemical markers. The study employs a randomized, placebo-controlled, crossover design to evaluate the efficacy of these supplements in enhancing overall health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Trouble falling asleep > 5 times a month (NHANES criteria)
* Body mass index 18.5-29.9 kg/m2
* Free of major chronic diseases or acute disorders
* Given written informed consent

Exclusion Criteria:

* History of dietary supplement use > 2 weeks before the study commences
* Abnormal values for lab clinical chemistry (> 2 SD)
* Unwillingness to return for follow-up analysis
* Participation in other clinical trials
* Moderate-to-heavy use of alcohol (> 3 drinks per week)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Total sleep time | Change from baseline total sleep time at 8 weeks
  Total sleep time measured with actigraph monitor

SECONDARY OUTCOMES:
Melatonin | Change from baseline serum melatonin at 8 weeks
  Level of serum melatonin in serum
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline PSQI at 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report tool used to assess sleep quality and disturbances. It consists of 19 items covering seven components: sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, daytime dysfunction, and use of sleep medications. Each component is scored from 0 to 3, with higher scores indicating worse sleep quality. The total score ranges from 0 to 21, where a score of 5 or higher suggests poor sleep quality. The PSQI is widely used in clinical and research settings to evaluate sleep health.

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Bioenergetics Lab at Faculty of Sport and PE, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in sleep medicine. Data will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Only qualified researchers with academic interest in sleep medicine